CLINICAL TRIAL: NCT01708941
Title: A Randomized Phase II Study of Ipilimumab at 3 mg/kg or 10 mg/kg Alone or in Combination With High Dose Interferon-Alpha in Advanced Melanoma
Brief Title: Ipilimumab With or Without High-Dose Recombinant Interferon Alfa-2b in Treating Patients With Stage III-IV Melanoma That Cannot Be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01932; NCI-2012-01932 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000741878; ECOG-E3611; E3611; E3611 (Other: ECOG-ACRIN Cancer Research Group); E3611 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Melanoma; Stage IIIA Cutaneous Melanoma AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; CTLA-4 Antigen; Introns; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A (higher dose ipilimumab, HDI) (Experimental): INDUCTION PHASE: Patients receive higher dose ipilimumab IV over 90 minutes once every 3 weeks for 4 doses and recombinant interferon alfa-2b IV over 20 minutes 5 days a week for 4 weeks and then SC 3 times weekly for 8 weeks.
  MAINTENANCE PHASE: Patients receive higher dose ipilimumab IV over 90 minutes once every 12 weeks for 4 doses beginning in week 24 and recombinant interferon alfa-2b SC 3 times weekly for 48 weeks.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Recombinant Interferon Alfa-2b
- Arm B (higher dose ipilimumab) (Experimental): INDUCTION PHASE: Patients receive higher dose ipilimumab IV over 90 minutes once every 3 weeks for 4 doses.
  MAINTENANCE PHASE: Patients receive higher dose ipilimumab IV over 90 minutes once every 12 weeks for 4 doses beginning in week 24.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis
- Arm C (lower dose ipilimumab + HDI) (Experimental): INDUCTION PHASE: Patients receive lower dose ipilimumab IV over 90 minutes once every 3 weeks for 4 doses and recombinant interferon alfa-2b IV over 20 minutes 5 days a week for 4 weeks and then SC 3 times weekly for 8 weeks.
  MAINTENANCE PHASE: Patients receive lower dose ipilimumab IV over 90 minutes once every 12 weeks for 4 doses beginning in week 24 and recombinant interferon alfa-2b SC 3 times weekly for 48 weeks.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Recombinant Interferon Alfa-2b
- Arm D (lower dose ipilimumab) (Experimental): INDUCTION PHASE: Patients receive lower dose ipilimumab IV over 90 minutes once every 3 weeks for 4 doses.
  MAINTENANCE PHASE: Patients receive lower dose ipilimumab IV over 90 minutes once every 12 weeks for 4 doses beginning in week 24.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Recombinant Interferon Alfa-2b — Given IV or SC
  Other Names: Alfatronol; Bioferon; Bioferon (TM); Glucoferon; Heberon Alfa; IFN alpha-2B; Interferon alfa 2b; Interferon Alfa-2B; Interferon Alpha-2b; Intron A; Sch 30500; Urifron; Viraferon
  Arms: Arm A (higher dose ipilimumab, HDI); Arm C (lower dose ipilimumab + HDI)

SUMMARY:
This randomized phase II trial studies how well ipilimumab with or without high-dose recombinant interferon alpha-2b works in treating patients with stage III-IV melanoma that cannot be removed by surgery. Monoclonal antibodies, such as ipilimumab, may block tumor growth by targeting certain cells. Recombinant interferon alfa-2b may interfere with the growth of tumor cells. It is not yet known whether ipilimumab is more effective with or without high-dose recombinant interferon alfa-2b in treating melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Test the hypothesis that the combination of ipilimumab and high-dose interferon-alpha 2b (HDI [recombinant interferon alfa-2b]) will improve progression free survival (PFS) of patients with advanced metastatic melanoma as compared to ipilimumab alone (across ipilimumab treatment status).

SECONDARY OBJECTIVES:

I. Test the hypothesis that the combination of ipilimumab and HDI will prove to be safe and tolerable.

II. Within the constraints of the sample size, attempt to test the hypotheses that (1) ipilimumab 10 mg/kg will lead to improved PFS in comparison to ipilimumab 3 mg/kg (across HDI treatment status); (2) the combination of ipilimumab and HDI will improve overall survival (OS) of patients with advanced metastatic melanoma as compared to ipilimumab alone (across ipilimumab treatment status) and (3) ipilimumab 10 mg/kg will lead to improved OS in comparison to ipilimumab 3 mg/kg (across HDI treatment status).

OUTLINE: Patients are randomized to 1 of 4 treatment arms.

ARM A:

INDUCTION PHASE: Patients receive higher dose ipilimumab intravenously (IV) over 90 minutes once every 3 weeks for 4 doses and recombinant interferon alfa-2b IV over 20 minutes 5 days a week for 4 weeks and then subcutaneously (SC) 3 times weekly for 8 weeks.

MAINTENANCE PHASE: Patients receive higher dose ipilimumab IV over 90 minutes once every 12 weeks for 4 doses beginning in week 24 and recombinant interferon alfa-2b SC 3 times weekly for 48 weeks.

ARM B:

INDUCTION PHASE: Patients receive higher dose ipilimumab IV over 90 minutes once every 3 weeks for 4 doses.

MAINTENANCE PHASE: Patients receive higher dose ipilimumab IV over 90 minutes once every 12 weeks for 4 doses beginning in week 24.

ARM C:

INDUCTION PHASE: Patients receive lower dose ipilimumab IV over 90 minutes once every 3 weeks for 4 doses and recombinant interferon alfa-2b IV over 20 minutes 5 days a week for 4 weeks and then SC 3 times weekly for 8 weeks.

MAINTENANCE PHASE: Patients receive lower dose ipilimumab IV over 90 minutes once every 12 weeks for 4 doses beginning in week 24 and recombinant interferon alfa-2b SC 3 times weekly for 48 weeks.

ARM D:

INDUCTION PHASE: Patients receive lower dose ipilimumab IV over 90 minutes once every 3 weeks for 4 doses.

MAINTENANCE PHASE: Patients receive lower dose ipilimumab IV over 90 minutes once every 12 weeks for 4 doses beginning in week 24.

In all arms, treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have unresectable stage III or stage IV melanoma, either initial presentation or recurrent, that is of cutaneous origin or unknown primary origin and that is histologically diagnosed
* No more than one prior systemic therapeutic regimen for unresectable stage III or stage IV melanoma; this includes chemotherapy, biologic therapy, biochemotherapy, or investigational treatment; this does not include any therapies given in the adjuvant setting; however, patients are excluded if they have a history of prior treatment for melanoma (either adjuvant or metastatic disease) with ipilimumab or other cytotoxic T-lymphocyte antigen 4 (CTLA-4) inhibitor, or prior interferon-alpha treatment for metastatic disease (history of adjuvant interferon-alpha is allowed); there should be a 4-week washout period between last treatment administration and initiation of study therapy
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Patients must not have other significant medical, surgical, or psychiatric conditions or require any medication or treatment that in the opinion of the investigator may interfere with compliance, make the administration of ipilimumab or HDI hazardous or obscure the interpretation of adverse events (AEs), such as a condition associated with frequent diarrhea; patients must not have an active infection requiring current treatment with parenteral antibiotics
* Patients must not have a history of inflammatory bowel disease or diverticulitis (history of diverticulosis is allowed)
* Patients who have other current malignancies are not eligible; patients with other malignancies are eligible if they have been continuously disease free for > 5 years prior to the time of randomization; one exception are patients treated with a curative intent and are continuously disease free for > 3 years; these patients would be considered eligible:

  * Patients with prior history at any time of any in situ cancer, lobular carcinoma of the breast in situ, cervical cancer in situ, atypical melanocytic hyperplasia or Clark I melanoma in situ are eligible
  * Patients with prior history of basal or squamous skin cancer are eligible
* Patients must not have autoimmune disorders or conditions of immunosuppression that require current ongoing treatment with systemic corticosteroids (or other systemic immunosuppressants), including oral steroids (e.g., prednisone, dexamethasone) or continuous use of topical steroid creams or ointments or ophthalmologic steroids; a history of occasional (but not continuous) use of steroid inhalers is allowed; replacement doses of steroids for patients with adrenal insufficiency are allowed; patients who discontinue use of these classes of medication for at least 2 weeks prior to randomization are eligible if, in the judgment of the treating physician investigator, the patient is not likely to require resumption of treatment with these classes of drugs during the study; exclusion from this study also includes patients with a history of symptomatic autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, Sjogren's syndrome, autoimmune vasculitis [e.g., Wegener's granulomatosis]); motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre syndrome and Myasthenia gravis); other central nervous system (CNS) autoimmune disease (e.g., poliomyelitis, multiple sclerosis); patients with autoimmune hypothyroid disease or type I diabetes on replacement treatment are eligible
* Due to the possible effect of treatment with ipilimumab on the immunologic response to infectious disease vaccines, patients must not have had any infectious disease vaccination (e.g, standard influenza, H1N1 influenza, pneumococcal, meningococcal, tetanus toxoid) within 4 weeks prior to randomization
* Women must not be pregnant or breast-feeding; all females of childbearing potential must have a blood test or urine study during screening to rule out pregnancy; NOTE: a woman of childbearing potential (WOCBP) is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months); for the purposes of this study, post-menopause is defined as:

  * Amenorrhea >= 24 consecutive months without another cause, or
  * For women with irregular menstrual periods and taking hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level >= 35 mIU/mL Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential; men of fathering potential and WOCBP must be using an adequate method of contraception or must abstain from sexual intercourse to avoid conception/pregnancy throughout the study and for up to 26 weeks after the last dose of ipilimumab or HDI in such a manner that the risk of pregnancy is minimized; men or WOCBP who are unwilling or unable to strictly follow this requirement are not eligible
* White blood cells (WBC) >= 3000/uL
* Absolute neutrophil count (ANC) >= 1500/uL
* Platelets >= 100 x 10^3/uL
* Hemoglobin >= 10 g/dL
* Serum creatinine =< 1.8 mg/dl
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN) for patients with liver metastases and =< 2.0 x ULN for patients without liver metastases
* Serum bilirubin < 2 x ULN for patients with liver metastases and =< 1.5 x ULN for patients without liver metastases, (except patients with Gilbert's syndrome, who must have a total bilirubin < 3.0 mg/dL)
* No active or chronic infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Patients must be free of brain metastasis by contrast-enhanced computed tomography (CT)/magnetic resonance imaging (MRI) scans within 4 weeks prior to enrollment; if known to have prior brain metastases, must not have evidence of active brain disease after definitive therapy (surgery, radiation therapy or stereotactic radiosurgery) on two successive MRI evaluations at least 3 months apart (one of which is =< 4 weeks prior to starting the study drugs)
* All sites of disease must be evaluated within 4 weeks prior to randomization; patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-01-18 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Tarhini, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (277):
- United States (277):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York Oncology Hematology PC - Albany Medical Center, Albany, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Summa Health System - Akron Campus, Akron, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ECOG-ACRIN member institutions between 1/18/2013 and 11/30/2015.
Groups:
- Arm A (Higher Dose Ipilimumab, HDI): INDUCTION PHASE: Patients receive higher dose ipilimumab IV over 90 minutes once every 3 weeks for 4 doses and recombinant interferon alfa-2b IV over 20 minutes 5 days a week for 4 weeks and then SC 3 times weekly for 8 weeks.
  MAINTENANCE PHASE: Patients receive higher dose ipilimumab IV over 90 minutes once every 12 weeks for 4 doses beginning in week 24 and recombinant interferon alfa-2b SC 3 times weekly for 48 weeks.
  Ipilimumab: Given IV
  Recombinant Interferon Alfa-2b: Given IV or SC
- Arm B (Higher Dose Ipilimumab): INDUCTION PHASE: Patients receive higher dose ipilimumab IV over 90 minutes once every 3 weeks for 4 doses.
  MAINTENANCE PHASE: Patients receive higher dose ipilimumab IV over 90 minutes once every 12 weeks for 4 doses beginning in week 24.
  Ipilimumab: Given IV
- Arm C (Lower Dose Ipilimumab + HDI): INDUCTION PHASE: Patients receive lower dose ipilimumab IV over 90 minutes once every 3 weeks for 4 doses and recombinant interferon alfa-2b IV over 20 minutes 5 days a week for 4 weeks and then SC 3 times weekly for 8 weeks.
  MAINTENANCE PHASE: Patients receive lower dose ipilimumab IV over 90 minutes once every 12 weeks for 4 doses beginning in week 24 and recombinant interferon alfa-2b SC 3 times weekly for 48 weeks.
  Ipilimumab: Given IV
  Recombinant Interferon Alfa-2b: Given IV or SC
- Arm D (Lower Dose Ipilimumab): INDUCTION PHASE: Patients receive lower dose ipilimumab IV over 90 minutes once every 3 weeks for 4 doses.
  MAINTENANCE PHASE: Patients receive lower dose ipilimumab IV over 90 minutes once every 12 weeks for 4 doses beginning in week 24.
  Ipilimumab: Given IV
Period: Overall Study
Arm/Group | Arm A (Higher Dose Ipilimumab, HDI) | Arm B (Higher Dose Ipilimumab) | Arm C (Lower Dose Ipilimumab + HDI) | Arm D (Lower Dose Ipilimumab)
Started | 21 | 23 | 22 | 22
Eligible and Started Treatment | 18 | 22 | 19 | 22
Completed | 3 | 5 | 3 | 4
Not Completed | 18 | 18 | 19 | 18
Not completed — Adverse Event | 4 | 6 | 1 | 0
Not completed — Death | 1 | 1 | 2 | 14
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 4
Not completed — Disease progression | 9 | 10 | 8 | 0
Not completed — Alternative therapy | 0 | 0 | 2 | 0
Not completed — Ineligible and never started treatment | 1 | 0 | 1 | 0
Not completed — Never started treatment | 2 | 1 | 0 | 0
Not completed — Ineligible | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Eligible patients who began treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Higher Dose Ipilimumab, HDI) | Arm B (Higher Dose Ipilimumab) | Arm C (Lower Dose Ipilimumab + HDI) | Arm D (Lower Dose Ipilimumab) | Total
Number analyzed (Participants) | 18 | 22 | 19 | 22 | 81
Age, Continuous [Median (Full Range); unit: years] | 60 [20 to 74] | 57 [27 to 83] | 65 [29 to 77] | 57 [26 to 73] | 58 [20 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 6 | 9 | 33
  Male | 8 | 14 | 13 | 13 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 16 | 22 | 18 | 22 | 78
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 18 | 22 | 18 | 21 | 79
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was defined as time from randomization to any documented disease progression or death from any cause, whichever occurred first (event), or censored at last date known alive.
Time Frame: Assessed every 3 months for two years, then every 6 months for 3 years, then every 12 months for up to 10 years
Population: Assessed among eligible patients who started treatment. The primary objective of the study is to compare PFS on the combination of ipilimumab + HDI (Arms A & C) versus ipilimumab alone (Arms B & D), across ipilimumab treatment status. Thus data across arms are combined.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Ipilimumab + HDI: INDUCTION PHASE: Patients receive ipilimumab IV over 90 minutes once every 3 weeks for 4 doses and recombinant interferon alfa-2b IV over 20 minutes 5 days a week for 4 weeks and then SC 3 times weekly for 8 weeks.
  MAINTENANCE PHASE: Patients receive higher dose ipilimumab IV over 90 minutes once every 12 weeks for 4 doses beginning in week 24 and recombinant interferon alfa-2b SC 3 times weekly for 48 weeks.
  Ipilimumab: Given IV
  Recombinant Interferon Alfa-2b: Given IV or SC
- Ipilimumab Alone: INDUCTION PHASE: Patients receive ipilimumab IV over 90 minutes once every 3 weeks for 4 doses.
  MAINTENANCE PHASE: Patients receive higher dose ipilimumab IV over 90 minutes once every 12 weeks for 4 doses beginning in week 24.
  Ipilimumab: Given IV
Arm/Group | Ipilimumab + HDI | Ipilimumab Alone
Number analyzed (Participants) | 37 | 44
months | 7.5 [5.1 to 11.0] | 4.4 [2.7 to 8.2]
Statistical Analysis 1: Comparison: Ipilimumab + HDI vs Ipilimumab Alone; The primary comparison was ipilimumab + HDI versus ipilimumab alone, across ipilimumab dose (Arms A & C versus Arms B & D); Test type: Superiority; p = 0.490, Log Rank

2. Secondary Outcome: Progression-free Survival
Description: as for outcome 1
Time Frame: Assessed every 3 months for two years, then every 6 months for 3 years, then every 12 months for up to 10 years
Population: Eligible patients who started treatment; PFS comparison of higher dose ipilimumab versus lower dose ipilimumab across HDI status (Arms A & B versus Arms C & D)
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Higher Dose Ipilimumab (With or Without HDI): INDUCTION PHASE: Patients receive higher dose ipilimumab IV over 90 minutes once every 3 weeks for 4 doses and recombinant interferon alfa-2b IV over 20 minutes 5 days a week for 4 weeks and then SC 3 times weekly for 8 weeks.
  MAINTENANCE PHASE: Patients receive higher dose ipilimumab IV over 90 minutes once every 12 weeks for 4 doses beginning in week 24 and recombinant interferon alfa-2b SC 3 times weekly for 48 weeks.
  Ipilimumab: Given IV
  Recombinant Interferon Alfa-2b: Given IV or SC
- Lower Dose Ipilimumab (With or Without HDI): INDUCTION PHASE: Patients receive lower dose ipilimumab IV over 90 minutes once every 3 weeks for 4 doses and recombinant interferon alfa-2b IV over 20 minutes 5 days a week for 4 weeks and then SC 3 times weekly for 8 weeks.
  MAINTENANCE PHASE: Patients receive lower dose ipilimumab IV over 90 minutes once every 12 weeks for 4 doses beginning in week 24 and recombinant interferon alfa-2b SC 3 times weekly for 48 weeks.
  Ipilimumab: Given IV
  Recombinant Interferon Alfa-2b: Given IV or SC
Arm/Group | Higher Dose Ipilimumab (With or Without HDI) | Lower Dose Ipilimumab (With or Without HDI)
Number analyzed (Participants) | 40 | 41
months | 6.5 [5.1 to 13.5] | 3.8 [2.6 to 7.5]
Statistical Analysis 1: Comparison: Higher Dose Ipilimumab (With or Without HDI) vs Lower Dose Ipilimumab (With or Without HDI); PFS comparison of higher dose ipilimumab versus lower dose ipilimumab (Arms A & B versus Arms C & D); Test type: Superiority; p = 0.144, Log Rank

3. Secondary Outcome: Overall Survival (OS)
Description: Time from randomization to death (event), or censored at last date known alive
Time Frame: Assessed every 3 months for two years, then every 6 months for 3 years, then every 12 months for up to 10 years
Population: Eligible patients who started treatment; OS comparison of ipilimumab + HDI versus ipilimumab alone, across ipilimumab doses (Arms A & C versus Arms B & D)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab + HDI | Ipilimumab Alone
Number analyzed (Participants) | 37 | 44
months | 20.1 [8.5 to 33.6] | 24.7 [12.6 to 35.7]
Statistical Analysis 1: Comparison: Ipilimumab + HDI vs Ipilimumab Alone; Test type: Superiority; p = 0.691, Log Rank

4. Secondary Outcome: Overall Survival
Description: Time from randomization to death (event), or censored at last date known alive.
Time Frame: Assessed every 3 months for two years, then every 6 months for 3 years, then every 12 months for up to 10 years
Population: Eligible patients who started treatment; OS comparison of higher dose ipilimumab versus lower dose ipilimumab across HDI status (Arms A & B versus Arms C & D)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Higher Dose Ipilimumab (With or Without HDI) | Lower Dose Ipilimumab (With or Without HDI)
Number analyzed (Participants) | 40 | 41
months | 20.1 [10.4 to 31.4] | 23.5 [11.7 to 35.7]
Statistical Analysis 1: Comparison: Higher Dose Ipilimumab (With or Without HDI) vs Lower Dose Ipilimumab (With or Without HDI); Comparison of higher dose ipilimumab versus lower dose ipilimumab across HDI status (Arms A & B versus Arms C & D); Test type: Superiority; p = 0.868, Log Rank

5. Other Pre Specified Outcome: Clinical Response Rate
Description: Defined as the number of complete responses and partial responses per RECIST version 1.1 divided by the total number of evaluable cases
Time Frame: Assessed every 12 weeks for 3 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Immune-related Response Rate Per Immune-related Response Criteria
Description: Defined as the number of complete and partial responses per immune-related response criteria (irRC) divided by the total number of evaluable patients
Time Frame: Assessed every 12 weeks for 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment
Description: Adverse events were assessed in all patients who started treatment, regardless of eligibility. There were two ineligible patients on Arm C who began treatment who are included in this population.
Arm/Group | Arm A (Higher Dose Ipilimumab, HDI) | Arm B (Higher Dose Ipilimumab) | Arm C (Lower Dose Ipilimumab + HDI) | Arm D (Lower Dose Ipilimumab)
All-Cause Mortality (participants affected / at risk) | 11/18 | 13/22 | 14/21 | 13/22
Serious Adverse Events (participants affected / at risk) | 17/18 | 12/22 | 16/21 | 10/22
Other Adverse Events (participants affected / at risk) | 18/18 | 21/22 | 20/21 | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Higher Dose Ipilimumab, HDI) (N=18) | Arm B (Higher Dose Ipilimumab) (N=22) | Arm C (Lower Dose Ipilimumab + HDI) (N=21) | Arm D (Lower Dose Ipilimumab) (N=22)
Anemia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 9 | 2 | 8 | 1
Flu like symptoms (General disorders) | 2 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0
Endocrine disorders - Other, specify (Endocrine disorders) | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Nausea (Gastrointestinal disorders) | 5 | 1 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Autoimmune disorder (Immune system disorders) | 0 | 0 | 0 | 1
Encephalitis infection (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 3 | 1 | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 2 | 4 | 0
CPK increased (Investigations) | 2 | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 2 | 0 | 2
Lymphocyte count decreased (Investigations) | 1 | 0 | 2 | 0
Neutrophil count decreased (Investigations) | 4 | 1 | 3 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0
Serum amylase increased (Investigations) | 2 | 0 | 0 | 0
Weight loss (Investigations) | 1 | 0 | 0 | 0
White blood cell decreased (Investigations) | 3 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 1
Eye disorders - Other, specify (Eye disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 1
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Higher Dose Ipilimumab, HDI) (N=18) | Arm B (Higher Dose Ipilimumab) (N=22) | Arm C (Lower Dose Ipilimumab + HDI) (N=21) | Arm D (Lower Dose Ipilimumab) (N=22)
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 10 | 1 | 10 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 8 | 2 | 13 | 0
Edema limbs (General disorders) | 1 | 1 | 1 | 0
Fatigue (General disorders) | 16 | 14 | 17 | 12
Fever (General disorders) | 11 | 3 | 14 | 0
Flu like symptoms (General disorders) | 2 | 1 | 2 | 0
Infusion related reaction (General disorders) | 1 | 1 | 1 | 0
Injection site reaction (General disorders) | 2 | 0 | 1 | 0
Localized edema (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 1 | 1
Pain (General disorders) | 1 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 14 | 7 | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 15 | 14 | 6 | 11
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 2 | 3 | 1 | 1
Hypothyroidism (Endocrine disorders) | 5 | 2 | 2 | 3
Endocrine disorders - Other, specify (Endocrine disorders) | 6 | 4 | 6 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 5 | 2 | 2
Colitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 4 | 3
Diarrhea (Gastrointestinal disorders) | 11 | 7 | 7 | 8
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 13 | 4 | 9 | 7
Vomiting (Gastrointestinal disorders) | 11 | 4 | 3 | 3
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 7 | 4 | 12 | 2
Alkaline phosphatase increased (Investigations) | 5 | 2 | 6 | 5
Aspartate aminotransferase increased (Investigations) | 14 | 3 | 13 | 2
Blood bilirubin increased (Investigations) | 2 | 0 | 2 | 0
Blood corticotrophin decreased (Investigations) | 1 | 0 | 0 | 0
CPK increased (Investigations) | 4 | 0 | 3 | 0
Creatinine increased (Investigations) | 2 | 0 | 1 | 1
GGT increased (Investigations) | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 8 | 3 | 3 | 3
Lymphocyte count decreased (Investigations) | 6 | 0 | 4 | 0
Lymphocyte count increased (Investigations) | 1 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 9 | 2 | 9 | 1
Platelet count decreased (Investigations) | 7 | 0 | 9 | 0
Serum amylase increased (Investigations) | 4 | 4 | 6 | 3
Weight loss (Investigations) | 7 | 3 | 6 | 2
White blood cell decreased (Investigations) | 11 | 0 | 10 | 0
Investigations - Other, specify (Investigations) | 3 | 6 | 6 | 4
Anorexia (Metabolism and nutrition disorders) | 14 | 5 | 13 | 3
Dehydration (Metabolism and nutrition disorders) | 5 | 1 | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 | 0 | 7 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 0 | 3 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2 | 4 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 7 | 0 | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5 | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 3 | 6 | 3
Concentration impairment (Nervous system disorders) | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 7 | 0 | 3 | 0
Dysgeusia (Nervous system disorders) | 5 | 0 | 8 | 0
Headache (Nervous system disorders) | 4 | 4 | 4 | 7
Paresthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 2 | 0
Blurred vision (Eye disorders) | 1 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 2
Eye disorders - Other, specify (Eye disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 3 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 2 | 0
Depression (Psychiatric disorders) | 3 | 0 | 4 | 0
Insomnia (Psychiatric disorders) | 3 | 2 | 3 | 0
Restlessness (Psychiatric disorders) | 2 | 0 | 0 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 1
Hypotension (Vascular disorders) | 2 | 0 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT01708941/Prot_SAP_000.pdf